CLINICAL TRIAL: NCT01529307
Title: A Phase I, Open-label Dose Escalation Study With Safety Expansion of TAS266 Administered by IV Infusion to Patients With Advanced Solid Tumors
Brief Title: First in Human Trial of TAS266 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTAS266X2101
Record Dates: First submitted 2012-02-01; First posted 2012-02-08 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2012-12

CONDITIONS: Advanced Solid Tumors
Keywords: Biologic,; solid tumors,; Death Receptor 5 agonist,; caspase-8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAS266 (Experimental)
  Interventions: Drug: TAS266

INTERVENTIONS:
Drug: TAS266 — TAS266 IV infusions given weekly

SUMMARY:
This study will assess safety, tolerability, maximum tolerated dose or recommended dose for expansion of TAS266 administered by IV infusion to patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of solid tumors
* 18 years or older
* ECOG performance status of 0, 1 or 2
* Adequate bone marrow, hepatic and renal function
* Obtained written informed consent

Exclusion Criteria:

* Patients with primary CNS tumor or CNS tumor involvement. However patients with CNS metastases may be allowed if certain conditions are met.
* Major surgery within 4 weeks before study treatment
* Prior anaphylactic or other severe infusion reactions to human immunoglobulin or antibody formulations
* Impaired cardiac functions
* Previous hepatitis viral infection such as hepatitis B or hepatitis C
* Diagnosis of HIV infection
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Frequency and characteristics of Dose limiting toxicities at each dose level | 2 years

SECONDARY OUTCOMES:
Type, frequency, and severity of AEs, changes in laboratory and clinical assessments | 2 years
TAS266 serum concentrations and PK parameters: Cmax, Tmax, AUC0-tlast, Tlast, T1/2 and accumulation ratio of TAS266 | 8 timepoints each for Cycles 1 and 2, prior to dosing on Day 1 of Cycles 3, 4, 5 and 6, at End of Treatment
  1 Treatment Cycle = 28 days,) assuming maximum 6 cycles of treatment
Presence and concentration of anti-TAS266 antibodies | 2 Years
Tumor response | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - H. Lee Moffitt Cancer Center/University of South Florida Moffitt SC, Tampa, Florida
  - South Texas Accelerated Research Therapeutics START, San Antonio, Texas
  - University of Utah / Huntsman Cancer Institute Huntsman UT, Salt Lake City, Utah

REFERENCES:
- See also: Results for CTAS266X2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=9663